CLINICAL TRIAL: NCT05028712
Title: Development of a Multi-sensory Rehabilitation Program for People With Ultra Low Vision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2087742
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Low Vision Blindness; Visual Impairment; Quality of Life; Functional Visual Loss
Keywords: ultra low vision rehabilitation; multi sensory; functional vision assessment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Information Training (Experimental)
  Interventions: Behavioral: Visual Information Training
- Multimodal Training (Experimental)
  Interventions: Behavioral: Multimodal training

INTERVENTIONS:
Behavioral: Visual Information Training — Participants in this arm will receive training to improve the use of residual vision to enhance functional performance.
  Arms: Visual Information Training
Behavioral: Multimodal training — Participants in this arm will receive training in integrating input from different senses to enhance functional performance.
  Arms: Multimodal Training

SUMMARY:
This research is aimed to address one of the big gaps in the current vision rehabilitation protocols for people with profound visual impairment by evaluating a multisensory approach. There are a growing number of clinical trials that recruit people with end-stage eye diseases and the rehabilitation plan following various treatments is not clear. It is important to address this in order to maximize the efficacy of such treatments and to improve the quality of life in people with profound visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* People with ultra low vision (visual acuity ≤20/1600)

Exclusion Criteria:

* <12 years of age
* dependent on sighted guide
* cognitive impairment

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in visual ability | Baseline, 1 month, 3 months, 6 months
  Change in visual ability as measured by the Ultra Low Vision Visual Function Questionnaire. The scale measures both visual ability (Person Measure) and difficulty (Item Measure) in people with ultra low vision. 150 items on a likert scale ranging from 1 impossible, to 4 not difficult. Using a Rasch-Andrich rating model, Person Measures range from -6 to +2.8 logits, Item Measures range from -3.3 to +3.0 logits. Higher scores indicating better outcome.

SECONDARY OUTCOMES:
Change in hand-eye coordination | Baseline, 1 month, 3 months, 6 months
  Change in hand eye coordination as assessed by a leap motion (Ultra Leap) sensor taped to a Virtual Reality headset to track hand eye coordination.
Change in hearing ability | Baseline, 1 month, 3 months, 6 months
  Change in hearing ability as assessed by iHEARtest device (earphones, computer application). The participant presses the space bar on their computer keyboard every time they hear a sound. The iHEARtest provides a Hearing Number™ in each ear on a scale from 1=profound impairment, to 5= no impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Arathy Kartha, PhD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY College of Optometry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided